CLINICAL TRIAL: NCT00616317
Title: Register for Pediatric Patients With Antiphospholipid Syndrome (APS): European Project Extended Internationally Study
Acronym: APS
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Ministry of Higher Education, Science and Technology, Solvenia (Other Government)
Responsible Party: Sponsor
Other Study IDs: 235519
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Antiphospholipid Syndrome
Keywords: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to gather information about causes and treatment of Antiphospholipid Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or younger at the onset of disease
* Presence of Vascular Thrombosis
* UC Davis patient
* Presence of at least one Laboratory criteria including: Anticardiolipin antibody, Anti-B glycoprotein-I antibody or Lupus anticoagulant in plasma

Exclusion Criteria:

* Infants born to mothers with APS
* Infants with congenital thrombophilia

Ages: 1 Minute to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric Nephrology Clinic at University of California, Davis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-09; Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Long term survival | 10 year

CONTACTS AND LOCATIONS:
Overall Officials: Lavjay Butani, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-registry-study-for-pediatric-patients-with-antiphospholipid-syndrome-the-immune-system-wrongly-attacks-normal-blood-proteins-905091/